CLINICAL TRIAL: NCT06558981
Title: The Role of Adjuvant Radiotherapy in High Risk Locally Advanced Differentiated Thyroid Cancer：a 1:1 Randomized Phase III Clinical Trial
Brief Title: Adjuvant Radiotherapy in High Risk Locally Advanced DTC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Yu Wang, Chief of Head and Neck Surgery, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARAD-TC
Record Dates: First submitted 2024-07-26; First posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy + RAI (Experimental): Patients in the experimental group would receive radiotherapy and RAI.
  Interventions: Radiation: Radiotherapy; Other: radioiodine treatment
- RAI (Active Comparator): Patients in the control group would receive RAI.
  Interventions: Other: radioiodine treatment

INTERVENTIONS:
Radiation: Radiotherapy — Ppatients would receive external radiation therapy within 6 weeks after surgery, using intensity-modulated radiation therapy (IMRT) or volume modulated radiation therapy (VMAT) techniques. RAI would be administered as standard care. The treatment window is within 6 months after surgery.
  Arms: Radiotherapy + RAI
Other: radioiodine treatment — RAI would be delivered based on the condition of residual lesions after surgery. The treatment window is within 6 months after surgery.

SUMMARY:
This study is a phase III randomized controlled clinical trial on the role of adjuvant radiotherapy in high-risk locally advanced differentiated thyroid cancer. Patients who meet the inclusion criteria were randomly assigned 1:1 to either the experimental group (adjuvant radiotherapy+RAI) or the control group (RAI), with LRFS as the primary endpoint of the study.

ELIGIBILITY:
Inclusion Criteria:

1. The patient voluntarily joined this study and signed an informed consent form;
2. Age: ≥ 14 years old,<80 years old, male or female not limited;
3. Histopathological diagnosis of differentiated thyroid cancer;
4. Surgical total or near total thyroidectomy;
5. The surgery did not achieve R0 resection, and R1/ R2 resection was performed. The volume of residual tumor in R2 resected patients is less than 2cm3;
6. The main organ functions are normal;
7. Good compliance and cooperation with follow-up.

Exclusion Criteria:

1. Previously received radiation therapy for the head and neck area;
2. Differentiated thyroid cancer with poorly differentiated, or undifferentiated components;
3. There is distant metastasis;
4. Previously received 131I treatment;
5. Previously received or currently receiving targeted therapy, immunotherapy, chemotherapy;
6. Within 5 years or simultaneously suffering from other active malignant tumors. Cured local tumors, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, can be included in the group;
7. Pregnant or lactating women;
8. Other physical illnesses that affect patients' ability to receive standard treatment;
9. According to the researchers' assessment, there may be other factors that could force the subjects to terminate the study, such as suffering from other serious illnesses (including mental illnesses) that require concurrent treatment, severe abnormal laboratory test values, family or social factors that may affect the safety of the subjects or the collection of experimental data;
10. Individuals with claustrophobia who are unable to undergo radiation therapy;
11. Patients deemed unsuitable for inclusion by other attending physicians.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2031-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Local-regional Recurrence Free Survival （LRFS） | 5 years after surgery
  The time from surgery to the occurrence of local-regional tumor recurrence based on the RECIST 1.1. The definition of local areas includes thyroid area, cervical I-VII lymph nodes, and retropharyngeal lymph nodes.

SECONDARY OUTCOMES:
Local-regional Recurrence Rate，LRR | 5 years after surgery
  The percentage of patients with local-regional recurrence in the total number of patients.
Progression Free Survival，PFS | 5 years after surgery
  The time from surgery to tumor progression, including local recurrence and distant metastasis.
Overall Survival，OS | 5 years after surgery
  The time from surgery to patient death.
Adverse Events，AE | 5 years after surgery
  The name of AE (based on NCI-CTCAE V5.0 criteria), severity, duration, and correlation with radiotherapy;
Quality of Life as assessed by QLQ-H&N35 | 5 years after surgery
  Patients in the experimental group were evaluated for QoL within 1 week before the start of radiotherapy, 1 week after the end of radiotherapy, 3 months after the end of radiotherapy, and 1, 3, and 5 years after surgery. The control group patients were evaluated for QoL at 1 month, 3 months, 1 year, 3 years, and 5 years after surgery. The QoL evaluation scale adopts the EORTC Quality of Life Measurement Scale QLQ-H&N35 (V1.0) .
Quality of Life as assessed by QLQ-C30 | 5 years after surgery
  Patients in the experimental group were evaluated for QoL within 1 week before the start of radiotherapy, 1 week after the end of radiotherapy, 3 months after the end of radiotherapy, and 1, 3, and 5 years after surgery. The control group patients were evaluated for QoL at 1 month, 3 months, 1 year, 3 years, and 5 years after surgery. The QoL evaluation scale adopts the EORTC Quality of Life Measurement Scale QLQ-C30 (V3.0) Chinese version.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Univeristy Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided